CLINICAL TRIAL: NCT05679986
Title: Early Neurological Deterioration in Recent Small Subcortical Infarction：a Prospective Study
Brief Title: Early Neurological Deterioration in Recent Small Subcortical Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yuan Gao (Other)
Responsible Party: Sponsor-Investigator, Yuan Gao, Clinical Professor, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Other Study IDs: 2022-KY-1334-002
Record Dates: First submitted 2022-12-25; First posted 2023-01-11 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Infarction; Subcortical Infarction; Deterioration, Clinical; Progression
Keywords: Early Neurological Deterioration; Recent Small Subcortical Infarction
MeSH Terms: conditions — Cerebral Infarction; Clinical Deterioration; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Recent small subcortical infarction within 72 hours from stroke onset to admission: Recent small subcortical infarction (RSSI) is defined as small deep infarctions in the territory of perforating arteries with maximum axial diameters (MAD) of less than 20 mm. In this study, RSSIs in the territories of lenticulostriate area, pons are enrolled.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Recent small subcortical infarction (RSSI) is defined as a small deep infarction in the territory of a perforating artery with maximum axial diameters (MAD) of less than 20 mm. Although RSSI is generally considered to be of a relatively favorable prognosis, about 13.5% to 43% of RSSI patients experience early neurological deterioration (END) in the acute phase, which often bring adverse effects on long-term outcomes. Although a number of risk factors for END have been identified previously, however, the risk factors of END and the underlying etiological mechanism are still ambiguous, and also the relevant intervention measures lack sufficient evidences, which is a thorny problem that clinicians have to face.

In this multicenter, large-sample prospective registry study, we ought to investigate the natural course of END in patients with RSSI. Exploring the risk factors and potential mechanism of its occurrence and development, and trying to establish a comprehensive predictive model for END that integrates multi-dimensional information including clinical symptom, demographic data, biochemical biomarker and image data, and so as to provide a valuable tool for clinical evaluation and early management. Simultaneously, our study will provide information for the design of therapeutic randomized controlled trials in the future.

DETAILED DESCRIPTION:
RSSI patients within 72 hours of stroke onset were prospectively and consecutively enrolled from Janu 2015 to June 2024. After enrollment, Clinical data will be collected using an online electronic case report Form (e-CRF) at baseline and follow-up. Baseline data including demographic, first blood pressure, past and family history, past medications use, pre-stroke modified Rankin Scale score (mRS), assessment of mRS and NIHSS score on admission were recorded. After admission, NIHSS score was evaluated twice a day by two certified physicians, who were blinded to the study. laboratory tests including routine blood/biochemistry/renal function, etc.) Transthoracic echocardiogram, 24-hour Holter and neuroimages data including brain MRI/MRA/CTA/DSA, etc. were all collected. During hospitalization, the drug therapy (antiplatelet/anticoagulation, lipid-lowering, glucose lowering, antihypertensive, etc.) were also recorded. Early neurological deteriorations (END) were monitored by two certified physicians, who were blinded to the imaging, and the primary outcome of our study was the occurrence of END, which was defined as any increase of ≥ 2 points in the total NIHSS score or ≥ 1 point on the motor items of the NIHSS within 7 days of hospital admission with blind evaluation. And any new cerebrovascular events confirmed during hospitalization were recorded. By face-to face or telephone interviews, we extended the follow up to 1 year for our secondary outcome including ①percentage of patients with favorable functional recovery, defined as an mRS ≤1; ②Percentage of patients with new vascular events, defined as any stroke (ischemic or hemorrhage); ③Percentage of patients with the new clinical vascular events (ischemic stroke/ hemorrhagic stroke/ TIA/ MI/ vascular death) as a cluster and evaluated individually. ④Severe bleeding incidence (GUSTO definition), including fatal bleeding and symptomatic intracranial hemorrhage; ⑤ Incidence of symptomatic and asymptomatic intracranial hemorrhagic events; ⑥All-cause mortality; ⑦cognitive function (MOCA/MMSE score). The outcomes will be assessed by the neurologists blinded to study images. The quality control of all data will be held by the central center.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Time from the last seen normal to enrollment ≤ 72 h.
3. Completion of brain MRI (T1/T2/Flair/DWI sequences at least). The lesion belonged to the territory of the penetrating artery( lenticulostriate area and pons) on the DWI sequence and at least one of the vascular examinations such as MRA, CTA or DSA was completed.

Exclusion Criteria:

1. Patients with low imaging quality affecting the evaluation of the data;
2. Vascular malformations, aneurysms, intracranial hemorrhagic diseases, brain abscesses, malignant space occupying lesions or other non-ischemic intracranial lesions;
3. Patients with combined malignancy, hematological disease and other systemic diseases with possible hypercoagulable state;
4. pre-stroke mRS ≥2 ;
5. END occurred before the completion of brain MRI after admission;
6. Acute endovascular treatment had been received or was planed to be done;
7. Pregnant or lactating women;
8. Participating in another ongoing study;
9. Refused to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prospectively enroll consecutive patients with acute RSSI within 72 hours of onset January 2015 to January 2024.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Early Neurological Deterioration | within 7 days after admission
  any increase of ≥ 2 points in the total NIHSS score or ≥ 1 point on the motor items of the NIHSS within 7 days after admission

SECONDARY OUTCOMES:
Percentage of patients with favorable functional recovery | 12 months
  mRS ≤1
Percentage of patients with new vascular events | 12 months
  any stroke (ischemic or hemorrhage)
Percentage of patients with new clinical vascular events | 12 months
  ischemic stroke/ hemorrhagic stroke/ TIA/ MI/ vascular death as a cluster and evaluated individually
Severe bleeding | 12 months
  Severe bleeding incidence (GUSTO definition),including fatal bleeding and symptomatic intracranial hemorrhage.
All-cause mortality | 12 months
  All-cause mortality
cognitive function | 12 months
  MOCA/MMSE score

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Gao, doctor, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT05679986/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT05679986/ICF_001.pdf